CLINICAL TRIAL: NCT02318238
Title: Comparison Between 6 Minute Walk Test, 6 Minute Step Test and 4 Metre Gait Speed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Doctor in Physiotherapy, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FT001
Record Dates: First submitted 2014-12-04; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Healthy; Children
Keywords: evaluation; exercise tolerance; healthy children; 6MWT
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 6 minute walking test (Active Comparator): walking during 6 minutes
  Interventions: Other: 6 minutes walking test
- 6 minute step test (Experimental): stepping during 6 minutes
  Interventions: Other: 6 minutes step test
- 4 meter gait speed (Experimental): walking as fast as possible on 4 meters
  Interventions: Other: 4 meters gait speed

INTERVENTIONS:
Other: 6 minutes walking test
  Other Names: walk during 6 minutes as fast as possible
  Arms: 6 minute walking test
Other: 6 minutes step test
  Other Names: up and down a step during 6 minutes as fast as possible
  Arms: 6 minute step test
Other: 4 meters gait speed
  Other Names: walk a four metre distance
  Arms: 4 meter gait speed

SUMMARY:
The purpose of this study is to find an alternative to the six minute walk test by validating six minute step test and four metre gait speed in healthy children. Both tests were previously validated in adults and are easier to achieve in non-hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* a lung disease
* an overweight
* an orthopedic disability which can slow down the subject during tests execution

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Walked distance | At 6 minutes
  The distance walked by subjects during a 6 minute walk test
Steps count | At 6 minutes
  Steps number raised and lowered by subject during a 6 minute step test
Time | at 1 minute
  Time to walk four metres
6MWT speed | at 6 minutes
  Subjects speed (number of metres/minute) during the 6 minute walk test
6MST speed | at 6 minutes
  Number of steps/minute during the 6 minute step test
4MGS speed | at 1 minute
  Number of metres/second during the four metre gait speed

SECONDARY OUTCOMES:
Dyspnea | at 6 minutes
  Dyspnea is measured by a visual analogue scale
Perceived exertion | at 6 minutes
  Percieve exertion is measured by a perceive exertion scale
Heart rate | at 6 minutes
  Heart rate was measured after each test
Oxygen saturation | at 6 minutes
  Oxygen saturation was measured after each test

CONTACTS AND LOCATIONS:
Overall Officials: Sophie De Wulf, Principal Investigator — UCL
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium